CLINICAL TRIAL: NCT00913939
Title: MRI-Guided HDR Brachytherapy for Prostate Cancer
Brief Title: High-Dose-Rate Brachytherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB 09-0026-C
Record Dates: First submitted 2009-06-02; First posted 2009-06-04 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Patients With Prostate Cancer
Keywords: Prostate Cancer; HDR Brachytherapy; Prostate Brachytherapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: Salvage After EBRT (Active Comparator): Patients with locally recurrent prostate cancer after radiotherapy will receive tumor-targeted salvage HDR brachytherapy. Arm 1 of the study will be coordinated and closely integrated with a separate concurrent study of MRI-guided prostate biopsy, which will be performed prior to accrual to Arm 1 of this trial (UHN 05-0641-C).
  Interventions: Procedure: MRI Guided Needles to deliver HDR Brachytherapy
- 2: Boost to EBRT (Active Comparator): Patients with locally advanced prostate cancer will receive a boost of prostate-targeted HDR brachytherapy during external beam radiotherapy.
  Interventions: Procedure: MRI Guided Needles to deliver HDR Brachytherapy

INTERVENTIONS:
Procedure: MRI Guided Needles to deliver HDR Brachytherapy — Patients in this arm will receive two fractions (treatments) of brachytherapy over 14 days (+/- 7 days).
  Arms: 1: Salvage After EBRT
Procedure: MRI Guided Needles to deliver HDR Brachytherapy — Patients in this arm will receive 2 fractions (treatments) of brachytherapy before the start of RT, and 4-5 weeks towards the end of EBRT.
  Arms: 2: Boost to EBRT

SUMMARY:
This pilot study initiates a research program testing the early technical and clinical performance of a novel procedure for MRI-guided high-dose-rate (HDR) prostate brachytherapy. Testing will proceed in two cohorts of patients. In Arm 1, patients with locally recurrent prostate cancer after radiotherapy will receive tumor-targeted salvage HDR brachytherapy. Arm 1 of the study will be coordinated and closely integrated with a separate concurrent study of MRI-guided prostate biopsy, which will be performed prior to accrual to Arm 1 of this trial (UHN 05-0641-C). In arm 2, patients with locally advanced prostate cancer will receive a boost of prostate-targeted HDR brachytherapy during external beam radiotherapy.

This technique will be prospectively evaluated in up to 100 patients. Preliminary data acquired in this pilot study will determine the technical limits of MRI guided HDR brachytherapy and will be critical for the judicious conduct of a subsequent phase II clinical trial.

This proposal is innovative in two fundamental ways: MRI-guidance, and specific tumor targeting for HDR brachytherapy. Successful completion of this study will further individualize local therapy, not only for the benefit of the proportion of cancer patients for whom initial radiotherapeutic interventions have failed, but also provide valuable technical and clinical validation that these novel image-guided (IG) approaches are clinically feasible and could be applied more broadly in prostate cancer therapy.

DETAILED DESCRIPTION:
Two hundred and nineteen thousand new cases of prostate cancer have been projected in the Unites States for 2007, with external beam radiotherapy (EBRT) constituting the mainstay of local therapy for an increasing proportion of newly diagnosed patients. Despite improvements in the delivery and reduction in associated toxicity of external beam radiotherapy, local persistence or recurrence of disease remains prevalent in 25-51% of patients. Local disease after EBRT is a risk factor for subsequent metastatic progression and prostate cancer-specific mortality, and is a cause of morbidity including hematuria, obstructive uropathy, and chronic pain. Given its prevalence, and the lack of satisfactory local salvage treatments, fear of prostate cancer recurrence has been shown to impose a substantial burden of suffering in patients.

Stereotactic needle placement under MRI-guidance enables two critical steps in tumor-targeted brachytherapy: 1) directly guiding brachytherapy catheters to sites of tumor recurrence, and 2) permitting treatment planning and delivery to be based on 3D MRI images. MRI-based HDR brachytherapy will precisely identify the location of brachytherapy catheters relative to the target volumes and adjacent normal structures at risk of radiation injury, obviating the need for invasive saturation (24-100) mapping biopsies.

This study will build the evidence supporting the concept of MRI-guidance and tumor-targeted HDR brachytherapy in the management of prostate cancer. This trial will strive to demonstrate improvements in technical performance under MRI-guidance, while exploring a novel paradigm of patient-specific modulation of dose intensity based on regions of tumor burden.

ELIGIBILITY:
Inclusion Criteria:

* Prior enrollment of UHN 05-0641-C or UHN 12-5015-C (Arm 1)
* Histological evidence of recurrent prostate adenocarcinoma (Arm 1)
* PSA doubling time > 6 months (Arm 1)
* High-risk localized prostate cancer (>T2 or G>7 or PSA>20) (Arm 2)
* Planned for EBRT + HDR boost (+/- hormone therapy) (Arm 2)
* ECOG 0 or 1
* Age > 18 years
* Informed consent: All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

Exclusion Criteria:

* Radiological evidence of regional or distant metastases
* Contraindications to MRI (Patient weighing >136kg (scanner weight limit), Patients with pacemakers, cerebral aneurysm clips, shrapnel injury, or implantable electronic devices not compatible with MRI)
* Bleeding diathesis and anti-coagulative therapy that cannot be temporarily ceased during brachytherapy
* Previous prostate brachytherapy
* Active hormonal therapy (Arm 1)

  ->50% of contiguous sextants involved with tumor (Arm 1)
* Previous pelvic radiotherapy (Arm 2)
* Contraindications to endorectal coil, surgically absent rectum, severe hemorrhoids or colorectal surgery.
* Latex Allergy
* Contraindications to conscious sedation, local anesthesia, or spinal/epidural anesthesia.
* IPSS >18
* Large TURP defect
* TURP within the past 6 months
* Prostate gland size >80cc
* History of Ulcerative Colitis, Crohn's Disease, Ataxia Telangiectasia, or SLE
* Other medical conditions deemed by the PI to make patient ineligible for MRI-guided Prostate HDR brachytherapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2009-05; Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
To determine if MRI-guided HDR brachytherapy is associated with favorable measures of technical performance. | 5 years

SECONDARY OUTCOMES:
determine if prostate targeted & MRI-guided HDR BT is associated with favorable preliminary measures of clinical performance as boost to EBRT;if tumor-targeted & MRI-guided HDR BT is associated with favorable preliminary measures of clinical performance | 5 years
determine dose-response relationships for salvage brachytherapy with a 20% escalation in dose. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Chung, MB ChB, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada